CLINICAL TRIAL: NCT06587412
Title: Radial Shock Waves Versus Focal Shock Waves in the Treatment of Lateral Epicondylalgia
Brief Title: Treatment of Lateral Epicondylalgia With Shock Waves
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Professor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEIM/2024/4/101
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Epicondylitis of the Elbow; Epicondylitis, Lateral
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Radial Shock Wave Treatment (Experimental): Patients assigned to this group will receive three sessions. During each session, 2000 pulses will be administered using a radial shock wave generator, with a pressure of 2.5 bars and a frequency of 8 Hz.
  Interventions: Other: Radial shock waves treatment
- Focal Shock Wave Treatment (Experimental): Patients assigned to this group will receive three sessions. During each session, 2000 pulses will be delivered by a focal shock wave generator, with an energy flux density of 0.2 mJ/mm² and a frequency of 4 Hz.
  Interventions: Other: Focal Shock Waves treatment
- Placebo Shock Waves (Placebo Comparator): Subjects in this group will receive a placebo treatment with very low energy settings, designed to simulate therapy without offering real therapeutic effects. This group will receive 20 pulses per session, with an energy flux density of 0.08 mJ/mm².
  Interventions: Other: shock waves placebo treatment

INTERVENTIONS:
Other: Radial shock waves treatment — Subjects in this group will receive radial shock waves
  Arms: Radial Shock Wave Treatment
Other: Focal Shock Waves treatment — Subjects in this group will receive focal shock waves
  Arms: Focal Shock Wave Treatment
Other: shock waves placebo treatment — Subjects in this group will receive a shock waves placebo treatment with very low energy settings
  Arms: Placebo Shock Waves

SUMMARY:
Lateral epicondylalgia (LET) is characterized by pain, decreased muscle strength of the wrist extensor muscles, and disability. Among the treatments proposed in the literature, both focal shockwave therapy and radial shockwave therapy have been considered effective in the management of this musculoskeletal disorder. The objective of this study is to compare the safety and effectiveness of these two shockwave applications on the signs and symptoms of subjects with lateral epicondylalgia. In this clinical trial, subjects will be evaluated for elbow pain using a Visual Analog Scale (VAS), grip strength using a handheld dynamometer, and degree of disability using the Patient-Rated Tennis Elbow Evaluation Questionnaire (PRTEE). A six-month follow-up will be performed.

Patients will be randomly divided into three groups. The first group will receive radial shock waves (rESWT), the second group will receive focal shock waves (fESWT), and the third group, which will act as a control, will receive a placebo treatment with very low energy parameters according to the literature.

Subjects will receive three sessions, one session per week.

ELIGIBILITY:
Inclusion Criteria:

* Pain in the lateral epicondyle >3 months
* Pain when performing resisted grip
* Positive Cozen test
* Positive Maudsley test

Exclusion Criteria:

* Pregnancy
* Systemic diseases (Fibromyalgia, Diabetes, Arthritis)
* Local infection or Cancer
* Recent treatments (Physiotherapy, Corticosteroids)-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Pain with Visual Analogue Scale (VAS) | Change from Baseline pain at 6 month
  The pain VAS is a unidimensional measure of pain intensity, used to record patients' pain progression. VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured where "0" on the far left is no pain and "10" on the far right is the worst pain possible.

SECONDARY OUTCOMES:
Grip strength | Change from Baseline pain at 6 month
  Grip strength is a measure of muscular strength or the maximum force/tension generated by one's forearm muscles. It will be recorded using a hand-held dynamometer. The subject is asked to exert grip strength until pain appears. It is measured in newtons.
Patient Rated Tennis Elbow Evaluation (PRTEE) | Change from Baseline pain at 6 month
  The PRTEE is a population specific 15-item questionnaire designed to measure forearm pain and disability associated with lateral epicondyle tendinopathy. 0% is the best and 100% is the worst disability outcome
The Global Rating of Change (GROC) | Change from Baseline pain at 6 month
  It's a scale that assesses whether the patient condition has gotten worse, better, or stayed the same and to quantify the magnitude of that change, typically following treatment.Subjects will make global ratings of changes regarding their level of well-being from their neck pain since the initial examination on a 15-point self-report scale (from -7 to 7), where -7 is the worst possible value and 7 is the best possible value.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Investigación Fisioterapia y Dolor, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No